CLINICAL TRIAL: NCT00447928
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Dose-Ranging Study of the OrthoDerm Transdermal Nitroglycerin Patch for Patients With Chronic Lateral Epicondylitis
Brief Title: Phase II Dose-Ranging Study of OrthoDerm Patch for Patients With Tennis Elbow
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cure Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orthoderm-1-001-06
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Tendonitis
Keywords: tendonitis; nitroglycerin; nitric oxide; lateral epicondylitis
MeSH Terms: conditions — Tendinopathy; Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: OrthoDerm transdermal nitroglycerin patch

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of the use of low-dose nitroglycerin transdermal patches to treat pain and function in chronic tennis elbow.

DETAILED DESCRIPTION:
Chronic tendonitis remains difficult to treat. Nitric oxide has been demonstrated to stimulate tenocytes to proliferate, differentiate and produce matrix components including collagen. Studies have demonstrated that nitroglycerin transdermal patches, which release nitric oxide, reduce pain and increase function in patients with chronic tendonitis. The purpose of the present study is to examine the efficacy of three dose levels of nitroglycerin, compared to placebo, in reducing pain and increasing function in patients with chronic (greater than three months' duration) lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* males >18 yr and < 70 yr
* BMI < 38
* chronic lateral epicondylitis (symptomatic > 3 mo)
* pain on provocation >/- 4 on 11 point scale

Exclusion Criteria:

* patients on other pain medications
* bilateral elbow pain
* any humerus elbow or forearm fracture or surgery
* signs of injury other than lateral epicondylitis
* any concomitant disease or pain of the upper extremity
* orthostatic hypotension
* patients taking MAO inhibitors, phosphodiesterase inhibitors, adrenergic agents
* pregnant or nursing women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164
Dates: Start 2007-04; Study Completion 2007-11

PRIMARY OUTCOMES:
pain-free grip strength

SECONDARY OUTCOMES:
pain at rest
pain on provocation
function

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD, PhD, Study Chair — Cure Therapeutics, Inc
Locations (1):
- to Be Determined, Warsaw, Poland

REFERENCES:
- [Derived] Paoloni JA, Murrell GA, Burch RM, Ang RY. Randomised, double-blind, placebo-controlled clinical trial of a new topical glyceryl trinitrate patch for chronic lateral epicondylosis. Br J Sports Med. 2009 Apr;43(4):299-302. doi: 10.1136/bjsm.2008.053108. Epub 2008 Oct 29. PMID 18971247